CLINICAL TRIAL: NCT02704364
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled, Parallel Group, Multiple Center Study to Evaluate the Safety, Tolerability, and Efficacy of NGM282 Administered for 12 Weeks in Patients With Primary Sclerosing Cholangitis
Brief Title: A Study of NGM282 in Patients With Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0106; 2015-003392-30 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-10 (Estimated); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-03

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NGM282 Dose 1 (Experimental): NGM282 Dose 1
  Interventions: Biological: NGM282
- NGM282 Dose 2 (Experimental): NGM282 Dose 2
  Interventions: Biological: NGM282
- Placebo (Active Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM282
  Arms: NGM282 Dose 1; NGM282 Dose 2
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and activity of NGM282 in patients with Primary Sclerosing Cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PSC

Exclusion Criteria:

* Clinically significant acute or chronic liver disease of an etiology other than PSC
* Secondary or IgG4 related sclerosing cholangitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Rossi, PharmD, Study Director — NGM Biopharmaceuticals, Inc
Locations (38):
- United States (26):
  - NGM Clinical Study Site 118, Sacramento, California
  - NGM Clinical Study Site 112, San Clemente, California
  - NGM Clinical Study Site 127, San Francisco, California
  - NGM Clinical Study Site 106, Aurora, Colorado
  - NGM Clinical Study Site 115, Washington D.C., District of Columbia
  - NGM Clinical Study Site 110, Gainesville, Florida
  - NGM Clinical Study Site 124, Lakewood Rch, Florida
  - NGM Clinical Study Site 105, Miami, Florida
  - NGM Clinical Study Site 109, Indianapolis, Indiana
  - NGM Clinical Study Site 104, Detroit, Michigan
  - NGM Clinical Study Site 102, Kansas City, Missouri
  - NGM Clinical Study Site 107, St Louis, Missouri
  - NGM Clinical Study Site 103, New York, New York
  - NGM Clinical Study Site 116, Durham, North Carolina
  - NGM Clinical Study Site 120, Cincinnati, Ohio
  - NGM Clinical Study Site 114, Nashville, Tennessee
  - NGM Clinical Study Site 113, Dallas, Texas
  - NGM Clinical Study Site 117, Dallas, Texas
  - NGM Clinical Study Site 119, Houston, Texas
  - NGM Clinical Study Site 125, Southlake, Texas
  - NGM Clinical Study Site 111, Charlottesville, Virginia
  - NGM Clinical Study Site 122, Newport News, Virginia
  - NGM Clinical Study Site 101, Norfolk, Virginia
  - NGM Clinical Study Site 121, Richmond, Virginia
  - NGM Clinical Study Site 108, Seattle, Washington
  - NGM Clinical Study Site 126, Seattle, Washington
- NGM Clinical Study Site 301, Paris, France
- Netherlands (6):
  - NGM Clinical Study Site 402, Amsterdam
  - NGM Clinical Study Site 407, Amsterdam
  - NGM Clinical Study Site 406, Leiden
  - NGM Clinical Study Site 401, Nijmegen
  - NGM Clinical Study Site 404, Rotterdam
  - NGM Clinical Study Site 405, Utrecht
- United Kingdom (5):
  - NGM Clinical Study Site 505, Birmingham
  - NGM Clinical Study Site 504, Liverpool
  - NGM Clinical Study Site 502, London
  - NGM Clinical Study Site 501, Newcastle
  - NGM Clinical Study Site 503, Norwich

REFERENCES:
- [Derived] Sanyal AJ, Ling L, Beuers U, DePaoli AM, Lieu HD, Harrison SA, Hirschfield GM. Potent suppression of hydrophobic bile acids by aldafermin, an FGF19 analogue, across metabolic and cholestatic liver diseases. JHEP Rep. 2021 Feb 19;3(3):100255. doi: 10.1016/j.jhepr.2021.100255. eCollection 2021 Jun. PMID 33898959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 62 participants who met all inclusion criteria and no exclusion criteria were randomized to receive treatment over a 12-week treatment period at 24 clinic sites in the United States, 5 sites in the United Kingdom, 5 sites in the Netherlands, and 1 site in France.
Groups:
- NGM282 1.0 mg: Participants who were randomized to NGM282 1.0 mg self-administered NGM282 as an subcutaneous (SC) injection to the abdomen daily, at approximately the same time each morning, over the 12-week treatment period.
- NGM282 3.0 mg: Participants who were randomized to NGM282 3.0 mg self-administered NGM282 as an subcutaneous (SC) injection to the abdomen daily, at approximately the same time each morning, over the 12-week treatment period.
- Placebo: Participants who were randomized to placebo self-administered placebo as an subcutaneous (SC) injection to the abdomen daily, at approximately the same time each morning, over the 12-week treatment period.
Period: Overall Study
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Started | 21 | 21 | 20
Completed | 19 | 18 | 19
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Noncompliance with study drug | 1 | 1 | 0
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics were assessed in the Randomized Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 20 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 17 | 20 | 19 | 56
  >=65 years | 4 | 0 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (15.9) | 40.2 (13.0) | 43.4 (12.4) | 43.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 8 | 24
  Male | 14 | 12 | 12 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 18 | 16 | 52
  Black or African American | 1 | 2 | 4 | 7
  Asian | 1 | 0 | 0 | 1
  Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Alkaline Phosphatase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in alkaline phosphatase levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in ALP was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: International units/Liter
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
International units/Liter | 25.6 (100.3) | -9.8 (101.3) | -0.6 (79.5)
Statistical Analysis 1: Comparison: NGM282 1.0 mg vs Placebo; Test type: Superiority; p = 0.434, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimate = -14.0, 95% CI 2-sided [-68.0 to 28.0], Standard Error of Mean 21.4
Statistical Analysis 2: Comparison: NGM282 3.0 mg vs Placebo; Test type: Superiority; p = 0.646, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimate = 13.0, 95% CI 2-sided [-41.0 to 71.0], Standard Error of Mean 25.0

2. Secondary Outcome: Mean Percent Change From Baseline in Alkaline Phosphatase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in alkaline phosphatase levels.
Time Frame: Baseline to Week 12
Population: Mean percent change from baseline in ALP was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
percent change | 7.1 (5.8) | -4.2 (5.9) | -3.4 (6.0)

3. Secondary Outcome: Mean Rate of Change in Alkaline Phosphatase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess rate of change in alkaline phosphatase levels. Serum levels of alkaline phosphatase was measured in a central laboratory using standard enzymatic method. The unit of measure is U/L.
Time Frame: Baseline to Week 12
Population: Mean rate of change in ALP was assessed in participants with available data in the Full Analysis Set .
Measure: Mean (Standard Error); unit: U/L/Week
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg
Number analyzed (Participants) | 21 | 19
U/L/Week
  Weeks 1 through 4 | -17.7 (6.4) | -2.2 (6.1)
  Weeks 5 through 12 | 11.9 (4.5) | -0.2 (2.2)

4. Secondary Outcome: Mean Change From Baseline in Aspartate Aminotransferase and Alanine Aminotransferase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in aspartate aminotransferase and alanine aminotransferase levels.
Time Frame: Baseline to Week 12
Population: Mean changes from baseline in aspartate aminotransferase and alanine aminotransferase were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: units/liter
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
units/liter
  Aspartate aminotransferase | -0.2 (7.0) | -30.9 (7.0) | -13.3 (7.1)
  Alanine aminotransferase | 8.5 (10.2) | -45.1 (10.4) | -12.1 (10.5)

5. Secondary Outcome: Mean Percent Change From Baseline in Aspartate Aminotransferase and Alanine Aminotransferase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in aspartate aminotransferase and alanine aminotransferase levels.
Time Frame: Baseline to Week 12
Population: Mean percent changes from baseline in aspartate aminotransferase and alanine aminotransferase were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
percent change
  Aspartate aminotransferase | 2.6 (7.8) | -25.5 (7.9) | -7.2 (8.0)
  Alanine aminotransferase | 7.2 (8.1) | -29.2 (8.2) | -6.1 (8.3)

6. Secondary Outcome: Mean Change From Baseline in Bilirubin (Direct and Total) in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in bilirubin (direct and total) levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in bilirubin (total and direct) was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: micromole/liter
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
micromole/liter
  Direct bilirubin | 9.14 (5.19) | 0.54 (5.30) | 0.55 (5.2)
  Total bilirubin | 9.78 (5.88) | 0.04 (6.01) | 0.83 (6.02)

7. Secondary Outcome: Mean Percent Change From Baseline in Bilirubin (Direct and Total) in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in bilirubin (direct and total) levels.
Time Frame: Baseline to Week 12
Population: Mean percent changes from baseline in bilirubin (total and direct) were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
percent change
  Direct bilirubin | 36.5 (16.7) | 5.7 (17.1) | 9.2 (17.1)
  Total bilirubin | 27.2 (17.9) | -3.6 (18.2) | 6.8 (18.2)

8. Secondary Outcome: Mean Change From Baseline in Gamma Glutamyl Transferase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in gamma glutamyl transferase levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in gamma glutamyl transferase was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: units/liter
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
units/liter | 156.6 (45.7) | -20.3 (46.3) | 4.6 (46.5)

9. Secondary Outcome: Mean Percent Change From Baseline in Gamma Glutamyl Transferase in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in gamma glutamyl transferase levels.
Time Frame: Baseline to Week 12
Population: Mean percent change from baseline in gamma glutamyl transferase was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 20
percent change | 20.9 (10.5) | 6.6 (10.6) | 7.5 (10.6)

10. Secondary Outcome: Mean Change From Baseline in Cholesterol Levels in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in cholesterol levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in cholesterol levels were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: millimole/liter
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 20
millimole/liter
  Total cholesterol | 0.14 (1.01) | 0.26 (1.10) | 0.15 (0.69)
  High-density lipoprotein | 0.04 (0.46) | -0.05 (0.50) | -0.06 (0.19)
  Low-density lipoprotein | 0.07 (0.85) | 0.30 (0.71) | 0.12 (0.54)
  Triglycerides | 0.01 (0.59) | -0.08 (0.37) | 0.10 (0.34)

11. Secondary Outcome: Mean Percent Change From Baseline in Cholesterol Levels in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in cholesterol levels.
Time Frame: Baseline to Week 12
Population: Mean percent change from baseline in cholesterol levels were assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 20
percent change
  Total cholesterol | 1.81 (16.45) | 5.67 (16.31) | 3.89 (12.17)
  High-density lipoprotein | 0.47 (28.94) | -0.36 (23.87) | -3.09 (10.42)
  Low-density lipoprotein | 1.36 (27.56) | 10.63 (19.62) | 6.18 (19.15)
  Triglycerides | 3.47 (45.71) | -5.81 (27.22) | 11.61 (33.32)

12. Secondary Outcome: Mean Change From Baseline in 25-Hydroxyvitamin D in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in 25-Hydroxyvitamin D levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in 25-Hydroxyvitamin D was assessed in the Full Analysis Set.
Measure: Mean (Standard Error); unit: nmol/Liter
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 20
nmol/Liter | 6.4 (33.9) | 1.1 (30.6) | 0.7 (21.7)

13. Secondary Outcome: Mean Percent Change From Baseline in 25-Hydroxyvitamin D in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in 25-Hydroxyvitamin D levels.
Time Frame: Baseline to Week 12
Population: Mean percent change from baseline in 25-Hydroxyvitamin D was assessed in the Full Analysis Set.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 20
percent change | 30.5 (97.3) | 17.0 (64.8) | 4.4 (41.6)

14. Secondary Outcome: Mean Change From Baseline in Prothrombin International Normalized Ratio in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in Prothrombin levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in Prothrombin was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: International normalized ratio
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 19
International normalized ratio | 0.03 (0.09) | 0.01 (0.07) | 0.00 (0.08)

15. Secondary Outcome: Mean Percent Change From Baseline in Prothrombin International Normalized Ratio in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in Prothrombin levels.
Time Frame: Baseline to Week 12
Population: Mean percent change from baseline in Prothrombin was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 20 | 19
percent change | 3.39 (8.02) | 0.65 (6.67) | 0.47 (6.75)

16. Secondary Outcome: Mean Change From Baseline in Calprotectin in Patients With Primary Sclerosing Cholangitis
Description: Blood samples were collected to assess changes in Calprotectin levels.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in Calprotectin was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: microgram/gram
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 14 | 9 | 16
microgram/gram | 353.4 (839.8) | 211.8 (585.8) | -10.3 (457.9)

17. Secondary Outcome: Mean Change From Baseline in Enhanced Liver Fibrosis Score in Patients With Primary Sclerosing Cholangitis
Description: Enhanced Liver Fibrosis (ELF) score is a non-invasive blood test derived from the measurement of hyaluronic acid (HA), amino terminal propeptide of type III procollagen (PIIINP), and tissue inhibitor of metalloprotease 1 (TIMP1) using a proprietary algorithm (Siemens). ELF score is a laboratory test, is unitless, and is used as a continuous variable. The minimal ELF score is zero, the maximal ELF score is unknown. The higher the ELF score, the worse the disease outcome.
  ELF is a score on a scale of severity assessment against biopsy-proven fibrosis. A score of <7.7 is none to mild, > 7.7-9.8 is moderate, > 9.8 is severe.
Time Frame: Baseline to Week 12
Population: Mean change from baseline in Enhanced Liver Fibrosis Score was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 20
units on a scale | -0.22 (0.64) | -0.26 (0.66) | 0.05 (0.52)

18. Secondary Outcome: Severity of Inflammatory Bowel Disease-Associated Intestinal Symptoms in Patients With Primary Sclerosing Cholangitis
Description: Severity of inflammatory bowel disease (IBD)-associated symptoms and acute cholangitis are summarized with number and percentage. The partial Mayo IBD scale assesses stool frequency, rectal bleeding, and there is a Physician's global assessment. Each section is summed and remission is defined as a total score of 0-1, mild disease 2-4, moderate disease 5-6, and severe disease 7-9. Higher total scores indicate more severe disease. The number of participants are being presented based on the severity of their IBD symptoms.
Time Frame: Baseline to Week 12
Population: Severity of inflammatory bowel disease-associated intestinal symptoms were assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
Number analyzed (Participants) | 21 | 21 | 20
Participants
  Remission | 12 | 13 | 17
  Mild disease | 8 | 8 | 3
  Moderate disease | 1 | 0 | 0
  Severe disease | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Day 1 up to Week 16.
Arm/Group | NGM282 1.0 mg | NGM282 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/21 | 2/21 | 0/20
Other Adverse Events (participants affected / at risk) | 17/21 | 20/21 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NGM282 1.0 mg (N=21) | NGM282 3.0 mg (N=21) | Placebo (N=20)
Bowel obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NGM282 1.0 mg (N=21) | NGM282 3.0 mg (N=21) | Placebo (N=20)
Abdominal cramps (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia aggravated (Gastrointestinal disorders) | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 0
Increased stool frequency (Gastrointestinal disorders) | 1 | 3 | 0
Loose stools (Gastrointestinal disorders) | 4 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 3
Nausea aggravated (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 3
Injection site erythema (General disorders) | 2 | 11 | 1
Injection site pain (General disorders) | 1 | 1 | 2
Malaise (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 4
Rhinitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 4 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 4 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT02704364/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT02704364/SAP_001.pdf